CLINICAL TRIAL: NCT04919811
Title: A Single-Arm, Open-Label, Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of Taletrectinib in Patients With Advanced or Metastatic ROS1 Positive NSCLC and Other Solid Tumors
Brief Title: Taletrectinib Phase 2 Global Study in ROS1 Positive NSCLC
Acronym: TRUST-II
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-106-G208
Expanded Access: NCT06841874 (No longer available)
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — taletrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Taletrectinib (Experimental): Single-arm trial whereby all consented, enrolled, eligible patients receive taletrectinib
  Interventions: Drug: Taletrectinib

INTERVENTIONS:
Drug: Taletrectinib — 400mg or 600mg QD
  Other Names: DS-6051b; AB-106

SUMMARY:
The main purpose of the study is to evaluate safety and efficacy of taletrectinib (also known as AB-106 or DS-6051b) monotherapy in the treatment of advanced NSCLC.

DETAILED DESCRIPTION:
This is a global Phase 2, multicenter, single-arm, open label study of taletrectinib in patients of NSCLC harboring with ROS1 fusion gene.

About 214 patients will be enrolled and divided into 5 cohorts, depending on past history of ROS1 TKI treatment.

Taletrectinib is administered once daily in 21-day cycles. Patients will continue with the treatment on taletrectinib until progression of disease as determined by the investigator.

The tumor response evaluation will be conducted on a regular basis until progression of disease. Long-term survival follow-up will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years (or ≥20 years as required by local regulations).
2. Histologically or cytologically confirmed diagnosis of locally advanced (including inoperable Stage IIIA or IIIB NSCLC) or metastatic NSCLC (Cohorts 1-3, 5) or other solid tumors including NSCLC patients ineligible for other cohorts (Cohort 4).
3. Evidence of ROS1 fusion by a validated assay as performed in Clinical Laboratory Improvement Amendments (CLIA)-certified or locally equivalent diagnostic laboratories. The molecular assays (i.e., Reverse Transcription Polymerase Chain Reaction [RT-PCR], Next-generation Sequencing [NGS]) are highly recommended.
4. Sufficient tumor tissue is required for patients in Cohort 1 and for TKI-naïve patients in Cohort 5 in order to perform confirmatory ROS1 fusion testing at the designated central laboratories. For patients in Cohort 1 and for TKI-naïve patients in Cohort 5, an archival tumor tissue specimen should be available and collected prior to enrollment. If archival tumor tissue is unavailable, then a fresh biopsy must be performed. Tumor tissue for patients in other cohorts is highly recommended, and tumor tissue obtained after progression on the most recent prior ROS1 TKI therapy in these cohorts is preferred. Cytology samples (e.g., pleural effusion cell pellets) may be acceptable for patients in Cohorts 2-4, and patients in Cohort 5 that received prior treatment with TKI(s) having ROS1 activity.
5. Patients with central nervous system (CNS) involvement, including leptomeningeal carcinomatosis, must be stable (either asymptomatic or previously treated and controlled are allowed:

   * Seizure prophylaxis is permitted with non-enzyme inducing anti-epileptic drugs (non-EIAEDs).
   * Corticosteroid treatment at a stable or decreasing dose within 7 days prior to the first dose of taletrectinib.

     * Whole brain radiation therapy (WBRT) must be completed at least 14 days and stereotactic radiotherapy, stereotactic radiosurgery, or gamma knife radiotherapy at least 7 days prior to enrollment; the patient must be clinically stable for 7 days according to investigator judgement prior to first dose of taletrectinib.
6. The patient can be either ROS1 TKI treatment naïve or treated with prior ROS1 TKI(s):

   o Cohort 1: Patients with locally advanced or metastatic ROS1-positive NSCLC. Systemic chemotherapy naïve or pretreated with 1 prior line of chemotherapy but never treated with any ROS1 TKI.

   o Cohort 2: Patients with locally advanced or metastatic ROS1-positive NSCLC. Prior treatment with 1 approved ROS1 TKI (crizotinib or entrectinib) and disease progression. The patient can be either chemotherapy naïve or has received 1 line of systemic chemotherapy for locally advanced or metastatic ROS1-positive NSCLC.
   * Cohort 3: Patients with locally advanced or metastatic ROS1-positive NSCLC. Prior treatment with ≥2 TKIs with ROS1 activity and disease progression. The patient can be either chemotherapy naïve or has received 1 line of systemic chemotherapy for locally advanced or metastatic ROS1-positive NSCLC, patients with known ROS1 resistant mutations are preferred.
   * Cohort 4: Patients with other ROS1-positive solid tumors, or NSCLC patients ineligible for Cohorts 1-3. Prior treatment with ≤3 TKIs with ROS1 activity. The patient can be either chemotherapy naïve or has received ≤2 lines of systemic chemotherapy for locally advanced or metastatic solid tumors.
   * Cohort 5: Patients with locally advanced or metastatic ROS1-positive NSCLC. The patient can be either chemotherapy naïve or has received ≤2 lines of systemic chemotherapy line of systemic chemotherapy for locally advanced or metastatic ROS1-positive NSCLC. ROS1-TKI-naïve or pretreated with TKI(s) having ROS1 activity.
7. At least 1 measurable disease per RECIST 1.1 as assessed by the investigator.
8. Eastern Cooperative Oncology Group Performance Status: 0 or 1.
9. Patient with a life expectancy ≥12 weeks based on the judgement of investigator.
10. Patients with adequate organ function meeting the following criteria:

    1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT): ≤3.0 × upper limit of normal (ULN) (or ≤5.0 × ULN, for patients with concurrent liver metastases)
    2. Serum total bilirubin: ≤1.5 × ULN (≤3.0 × ULN for patients with Gilbert syndrome or if liver function abnormalities are due to underlying malignancy)
    3. Absolute neutrophil count: ≥1,500/μL
    4. Platelet count: ≥100,000/μL
    5. Hemoglobin: ≥9.0 g/dL
    6. Serum creatinine ≤1.5 × ULN and estimated creatinine clearance (CLcr) ≥45 mL/min as calculated using the method standard for the institution (e.g., Cockcroft - Gault Equation)
11. Males and/or females who meet any of the following criteria:

    a. For males (irrespective of surgical sterilization [vasectomy]): agree to use effective contraception methods during the study intervention period and for at least 90 days after the last dose of investigational drug or agree with complete abstinence.

    b. Females without menses for at least 1 year prior to screening or documented to be surgically sterilized. Women of childbearing potential (WOCBP) must agree to use two concurrent highly effective methods of contraception or agree with complete abstinence from sexual intercourse since the informed consent until 45 days after the last dose of investigational drug. Usage of hormonotherapy for contraception should be recorded as well.
12. For all females of childbearing potential, a negative pregnancy test must be obtained within 7 days before starting study treatment. Female patients of non childbearing potential must meet at least 1 of the following criteria:

    ○ Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed with a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state.

    ○ Have undergone a documented hysterectomy and/or bilateral oophorectomy.

    ○ Have medically confirmed ovarian failure. All other female patients (including female patients with tubal ligations) are considered to be of childbearing potential.
13. The patient is willing and capable to give written informed consent.
14. The patient is willing and capable to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
15. The patient is willing and capable to comply with study site's COVID-19 policies.

Exclusion Criteria

1. Treatment with small molecule anticancer therapy including other investigational agents or cytotoxic systemic anticancer therapy within 2 weeks (or 5 half-lives of the compound, whichever is shorter) prior to the first dose of taletrectinib; or treatment with monoclonal antibodies, including immune checkpoint inhibitors within 4 weeks before the first dose of taletrectinib.
2. Major surgical procedure, open biopsy, or significant traumatic injury ≤4 weeks before the first dose of taletrectinib.

   Note: Placement of vascular access device is not considered major surgery. Other minor surgical procedures, such as catheter placement or minimally invasive biopsy, are allowed.
3. Radiation outside the chest and brain <7 days prior to C1D1.
4. Have been diagnosed with another primary malignancy other than NSCLC except for adequately treated non-melanoma skin cancer or cervical cancer in situ; definitively treated non-metastatic prostate cancer; or patients with another primary malignancy who are definitively relapse-free with at least 3 years elapsed since the diagnosis of the other primary malignancy.
5. Adverse events due to prior therapy are unresolved to ≤ CTCAE Grade 1 or has not returned to baseline, by the first dose of taletrectinib except for AEs not constituting a safety risk to the patient based on the judgment of investigators.
6. Patients with untreated spinal cord compression caused by tumor and/or cancerous meningitis.
7. History or evidence of interstitial fibrosis, interstitial lung disease or drug-induced pneumonitis (Excluding clinically insignificant or asymptomatic post radiation pneumonitis).
8. Any gastrointestinal disorders that may affect absorption of oral medications.

1. 9. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV), hepatitis C virus (HCV), or severe acute respiratory syndrome coronavirus 2 (SARS CoV 2), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness. Note that the following are permitted:

○ Patients treated for hepatitis C (HCV) or HIV with no detectable viral load; for at least 1 month prior to the first dose of taletrectinib.

Note: caution with drug drug interactions of concomitant anti HIV agents and CYP3A substrates.

○ Patients with known hepatitis B (HBV) infections:

* With past or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of hepatitis B surface antigen [HBsAg]); or
* With inactive HBV carrier state (defined as HBsAg positive, with normal ALT, and HBV DNA <2,000 IU/mL or <10,000 copies/mL).

Note: Please consider that, for patients in an inactive HBV carrier state or with a resolved HBV infection, there may be a risk of HBV reactivation, and anti HBV prophylaxis should be considered.

10. Clinically significant cardiovascular diseases within 3 months prior to the first dose of taletrectinib: myocardial infarction, severe/unstable angina, coronary/peripheral endovascular treatment, heart failure or cerebrovascular disorder including transient ischemic attack.

11. Ongoing cardiac dysrhythmias of ≥ CTCAE Grade 2, uncontrolled atrial fibrillation of any grade, or QT interval corrected for heart rate by Fredericia's formula (QTcF) >470 milliseconds, or symptomatic bradycardia <45 beats per minute; patient has family or medical history of long QT syndrome.

12. Pregnancy or lactation/breastfeeding. 13. Use of food or drugs that are known potent cytochrome P450 3A4/5 (CYP3A4/5) inhibitors or inducers or P-glycoprotein inhibitors or inducers within 14 days prior to the first dose of study treatment and while on treatment.

14. Administration of agents with potential QT interval prolonging effect within 14 days prior to first dose of study treatment and while on treatment.

15. Patients with other severe medical or mental diseases in whom the risk is increased by participation to the study or treatment with study treatment in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by independent radiology review committee (IRC) | Up to 4 years
  Confirmed ORR according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 assessed by an independent radiology review committee (IRC)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 4 years
  PFS according to RECIST 1.1 assessed by IRC
Objective response rate (ORR) assessed by investigators | Up to 4 years
  ORR according to RECIST 1.1 assessed by investigators
Safety and tolerability of taletrectinib | Up to 4 years
  Incidence of Adverse events (AEs), incidence of laboratory abnormalities, incidence of abnormal vital signs, abnormal ECG and abnormal ophthalmologic findings
Pharmacokinetic (PK) profile of taletrectinib | Up to 4 years
  Maximum Plasma Concentration (Cmax) of taletrectinib

OTHER OUTCOMES:
Intracranial progression-free survival (IC-PFS) | Up to 4 years
  Confirmed IC-PFS per Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria
Intracranial objective response rate (IC-ORR) | Up to 4 years
  Confirmed IC-ORR per RANO-BM criteria

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, MD, PhD, Study Director — Nuvation Bio Inc.
Locations (77):
- United States (20):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - The Oncology Institute of Hope and Innovation, Glendale, California
  - Moores Cancer Center at UC San Diego, La Jolla, California
  - Keck Medicine of University of Southern California, Los Angeles, California
  - UCI Medical Center, Orange, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - SCRI - Florida Cancer Specialists South, Fort Meyers, Florida
  - Memorial Cancer Institute at Memorial Hospital East, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - SCRI - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - Mayo Clinic, Rochester, Minnesota
  - Center for Cancer Research, Brick, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, P.A., Dallas, Texas
  - Renovatio Clinical, El Paso, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre Research Institute, Montreal, Quebec
- China (8):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Chengdu
  - Shandong Cancer Hospital, Jinan
  - Wuhan Union Hospital, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- France (10):
  - CHU Lyon - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Bron
  - CHU Grenoble Alpes- Hospital Michallon, La Tronche
  - Centre Léon Bérard, Lyon 08
  - Centre d'Essais Précoces de Cancerologie de Marseille, Marseille
  - APHP- Hôpital Europeen Georges Pompidou (HEGP), Paris
  - CHU de Poitiers Pole regional, Poitiers
  - Institut Jean Godinot, Reims
  - CHU Rennes - Hospital Pontchaillou, Rennes
  - Institut De Cancérologie De L'ouest, Saint-Herblain
  - Institut Gustave Roussy, Saint-Herblain
- Italy (9):
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico, Bari
  - Humanitas Istituto Clinico Catanese, Misterbinanoco, Catania
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - AOU Cagliari- P.O. Policlinico Universitario Duilio Casula, Monserrato
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania, Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (8):
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Cancer Center Hospital East, Kashiwa
  - Sendai Kousei Hospital, Miyagi
  - Aichi Cancer Center Hospital, Nagoya
  - Kindai University Hospital, Osaka
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (3):
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Med-Polonia Sp. z o.o., Poznan
  - MICS Centrum Medyczne Toruńa, Torun
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Pusan National University Yangsan Hospital, Gyeongsang
  - Chonnam National University Hwasun Hospital, Hwasun
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (12):
  - Clinica Mi Tres Torres, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia IVO, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Perol M, Li W, Pennell NA, Liu G, Ohe Y, De Braud F, Nagasaka M, Felip E, Xiong A, Zhang Y, Fan H, Wang X, Li S, Lai RK, Ran F, Zhang X, Chen W, Bazhenova L, Zhou C. Taletrectinib in ROS1+ Non-Small Cell Lung Cancer: TRUST. J Clin Oncol. 2025 Jun;43(16):1920-1929. doi: 10.1200/JCO-25-00275. Epub 2025 Apr 3. PMID 40179330
- [Derived] Nagasaka M, Ohe Y, Zhou C, Choi CM, Yang N, Liu G, Felip E, Perol M, Besse B, Nieva J, Raez L, Pennell NA, Dimou A, Marinis F, Ciardiello F, Seto T, Hu Z, Pan M, Wang W, Li S, Ou SI. TRUST-II: a global phase II study of taletrectinib in ROS1-positive non-small-cell lung cancer and other solid tumors. Future Oncol. 2023 Jan;19(2):123-135. doi: 10.2217/fon-2022-1059. Epub 2023 Mar 6. PMID 36877099